CLINICAL TRIAL: NCT07282821
Title: Bempedoic Acid Therapy for Polycystic Kidney Disease (BEAT-PKD) Randomized Clinical Trial
Brief Title: Bempedoic Acid Therapy for Polycystic Kidney Disease
Acronym: BEAT-PKD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kenneth Hallows (Other)
Collaborators: University of Maryland, Baltimore County (Other); Tufts Medical Center (Other); University of Pittsburgh (Other); University of Southern California (Other); Biomedical Research Institute of New Mexico (Other)
Responsible Party: Sponsor-Investigator, Kenneth Hallows, Patrick Professor of Medicine and Network Division Chief of Nephrology, University of Vermont
Organization: University of Vermont (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00003795; HT94252510293 (Other Grant/Funding Number: U.S. Department of Defense)
Record Dates: First submitted 2025-12-05; First posted 2025-12-15 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: ADPKD (Autosomal Dominant Polycystic Kidney Disease)
Keywords: ADPKD; bempedoic acid; AMPK; ACLY; height-adjusted total kidney volume; biomarkers; MRI; urine; metabolism; tolvaptan
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Over-encapsulated bempedoic acid 180 mg p.o. once daily (Active Comparator)
  Interventions: Drug: Bempedoic Acid 180 MG Oral Tablet
- Matching over-encapsulated placebo pill given p.o. once daily (Placebo Comparator)
  Interventions: Drug: Placebo Capsule(s)

INTERVENTIONS:
Drug: Bempedoic Acid 180 MG Oral Tablet — Over-encapsulated active study drug
  Other Names: Nexletol
  Arms: Over-encapsulated bempedoic acid 180 mg p.o. once daily
Drug: Placebo Capsule(s) — Over-encapsulated placebo pill
  Arms: Matching over-encapsulated placebo pill given p.o. once daily

SUMMARY:
Autosomal dominant polycystic kidney disease (ADPKD), the most commonly inherited kidney disease, is characterized by the development of cysts in the kidney that impair function. Of those affected, half will progress to end-stage kidney disease by age 60, requiring dialysis or kidney transplant. To date, no effective and safe therapies exist for this deadly disease. Tolvaptan (Tol), the only FDA-approved drug for treatment of ADPKD, has some benefit in slowing kidney disease progression, but Tol causes frequent urination and thirst and also injures the liver in a small number of patients. The investigators' goal, therefore, is to develop new strategies to treat ADPKD that are safe and tolerable.

The development of cysts in ADPKD patients results from two main cellular processes. The first is cell growth with an increase in the number of kidney cells that make up the outer surface of the cyst. The second is an increase in fluid secretion into the cysts that develop. The investigators have shown that an enzyme, AMP-activated protein kinase (AMPK), when activated can inhibit both of those processes. Moreover, genetic mutations that cause ADPKD may alter the energy metabolism of the cell, which in turn inhibits AMPK activity. Bempedoic acid (BA), a medication that is FDA-approved for the treatment of individuals with high cholesterol and has a good safety record, activates AMPK. In addition to activating AMPK, BA inhibits a second enzyme called ATP-citrate lyase (ACLY), which is involved in cholesterol synthesis. ACLY has received growing attention as a novel target for cancer treatment. ACLY inhibition blocks increases of cell numbers by inhibiting the lipid synthesis that is required for creation of new cell membranes. This study will test whether targeting these pathways through treatment with BA will help reverse dysfunctional metabolism in individuals with ADPKD and slow disease progression.

The investigators will test this using a phase 2 clinical trial in which 120 individuals with rapidly progressive ADPKD and an estimated glomerular filtration rate of 35 or greater will be treated with either BA or placebo (inactive look-alike pill) for two years. Participants on or off a stable dose of Tol will be included in the study. Participants will be recruited from the U. of Vermont, U. of Maryland, and Tufts University, which have active PKD clinics and are recognized by the PKD Foundation as Centers of Excellence. Through follow-up visits and lab work, the investigators will assess the safety and tolerability of BA in the participants as the primary outcomes. The secondary goals are to assess preliminary efficacy and effects of BA on quality of life in study participants. The growth of cysts results in increased volume or size of the kidneys and liver. Total and cyst volumes of the kidney and liver and visceral abdominal fat content via magnetic resonance imaging (MRI) will be measured to gauge the effectiveness of this drug. The investigators also predict that proteins and small molecules involved in regulating cell energy metabolism, inflammation, and injury, as well as proteins directly involved in AMPK and ACLY function, will be altered in ADPKD patients. Levels of these proteins and small molecules may then subsequently change with BA therapy. Exploratory, mechanistic goals of this study are to identify prognostic and predictive urinary biomarkers in study participants. Successful completion of this study would have a significant impact on individuals with ADPKD by laying the groundwork for a new treatment strategy as well as by providing a new way to help guide treatment decisions.

In summary, the goals of this phase 2 randomized, double-blind, placebo-controlled clinical trial are to test the safety, tolerability and preliminary efficacy of the drug bempedoic acid, FDA-approved to lower cholesterol, when used in ADPKD patients.

DETAILED DESCRIPTION:
Background and Rationale: Autosomal Dominant Polycystic Kidney Disease (ADPKD) is the most common monogenic kidney disease affecting ~1:700 individuals with half of patients progressing to end-stage kidney disease by age 60. ADPKD is characterized by excessive epithelial cell proliferation and cAMP-dependent luminal fluid secretion that manifests as progressive cyst development. There is growing recognition that metabolic derangements occur in ADPKD cells contributing to cyst formation and expansion, including increased glycolysis, impaired mitochondrial fatty acid oxidation, and reduced activity of the metabolic sensor AMP-activated protein kinase (AMPK). Tolvaptan (Tol), the only FDA-approved drug for ADPKD, modestly slows disease progression in patients but has dose-dependent side effects limiting its tolerability, including polyuria and thirst, and rare hepatotoxicity, which requires close liver function test monitoring. New therapeutic strategies are greatly needed for ADPKD patients, especially ones that target complementary signaling pathways that may afford additivity in slowing disease progression when used together with Tol and may permit lower Tol dosing in patients. Recent preclinical work suggests that bempedoic acid (BA) may serve as an exciting new therapy for ADPKD in this regard. BA is an ATP-citrate lyase (ACLY) inhibitor FDA-approved to treat hypercholesterolemia. BA is a pro-drug that gets activated only in kidney and liver, the main organs affected in ADPKD, and catalyzes a key step in fatty acid and sterol synthesis important for cell growth and proliferation. BA also directly activates AMPK and promotes mitochondrial oxidative metabolism. Together, these effects target key dysregulated pathways in ADPKD and support the potential of this drug for the treatment of ADPKD. In preclinical studies BA treatment inhibited cyst growth and improved mitochondrial health in model ADPKD kidney cells and mice. Importantly, BA treatment appears to be safe and well tolerated in patients with mild-moderate CKD with no dose adjustment, although its use has never been studied specifically in ADPKD patients.

Hypothesis/Objectives: The investigators hypothesize that BA will be safe and tolerable in ADPKD patients and that repurposing BA for use in these patients will be beneficial in improving ADPKD disease features, both with and without concurrent Tol use. In Specific Aim 1 they will perform a randomized, placebo-controlled, double-blind, phase 2, multicenter clinical trial that will evaluate the safety, tolerability, quality of life, and preliminary efficacy of BA for 120 participants with ADPKD who are at high risk for rapid progression, either with or without concomitant Tol therapy, over a two-year period. Longitudinal changes in estimated GFR (eGFR), height-adjusted total kidney and liver volumes (htTKV and htTLV), kidney and liver cyst volumes (KCV and LCV), visceral abdominal fat, and urinary biomarkers will be assessed. In Specific Aim 2 the investigators will perform exploratory analyses and identification of prognostic and predictive urinary biomarkers related to disease severity and the expected metabolic effects of BA both before and after initiation of the study drug to evaluate potentially relevant biomarkers that correlate with ADPKD disease severity and response to BA.

Study Design: The investigators will perform a pilot-level, double-blind, phase 2, parallel-group, placebo-controlled multicenter clinical trial to evaluate BA in ADPKD patients over a two-year period. Each arm will consist of approximately 60 ADPKD patients who are at risk for rapid disease progression and may be either on or off tolvaptan, recruited from three geographically and ethnically diverse patient populations at Tufts U., U. Maryland, and U. Vermont. It is anticipated that each clinical site will recruit 40 participants who will be randomized in a 1:1 ratio to receive either placebo or BA (180 mg oral daily). For the primary endpoints, the study will evaluate safety, as defined by all and targeted adverse events (e.g., hyperuricemia/gout and liver transaminitis). Tolerability will be assessed by the % participants still taking study drug at 24 months and % adherence by pill counting, as well as the % participants who answer 'yes' to the question of whether they could tolerate taking the study drug for the rest of their lives. For the quality of life secondary endpoint, health-related quality of life metrics, including pain, discomfort, fatigue, emotional distress, and impaired mobility will be assessed via validated ADPKD questionnaires. For the secondary endpoint of preliminary efficacy, the investigators will estimate the effect of BA on htTKV, KCV, htTLV, LCV, and visceral abdominal fat by MRI at 0, 12, and 24 months during treatment, as well as estimated glomerular filtration rate (eGFR) by CKD-Epi and cystatin C equations with each visit. Clinical lab measurements will be performed at baseline prior to initiation of the study drug, at 2 weeks, 6 weeks, and 3 months, and then every 3 months thereafter for a total of 2 years. Patient surveys will be performed and urine will be collected from participants at each in-person study visit (occurring at baseline, 3, 6, 12, 18, and 24 months) to measure targeted urinary metabolic and other disease biomarkers that may correlate with ADPKD disease severity and response to BA. Inclusion criteria will include ADPKD patients aged 18-60 years, at risk for rapid disease progression with Mayo Imaging Classifications (MIC) 1C-1E or MIC 1B with defined eGFR decline >3 ml/min/yr, eGFR ≥35 ml/min, and English-speaking. Participants will be stratified by Tol use (stable Tol dose for >3 months prior to baseline visit). Exclusion criteria will include proteinuria >500 mg/day, current BA use, diabetes, known unstable cerebral aneurysm, active coronary artery disease, systemic kidney-impacting diseases, pregnancy or lactation, and implanted ferromagnetic objects.

Clinical Impact: Successful completion of this study could have a significant clinical impact, as it will provide the necessary foundation for a larger, phase 3 study to test BA efficacy in ADPKD patients. Given the established safety record and preclinical data showing the effects of BA in the disease process, it is expected that BA could alter clinical practice. Moreover, identification of biomarkers for disease severity and therapeutic response would significantly improve the management of ADPKD patients.

ELIGIBILITY:
Inclusion Criteria:

* ADPKD patients as defined by Pei-Ravine criteria
* Age 18-60 years
* Mayo Imaging Classifications (MIC) 1C-1E or MIC 1B with defined eGFR decline >3 ml/min/1.73m2/yr (estimated from serum creatinine using the CKD-Epi equation)
* Estimated glomerular filtration rate (eGFR) ≥35 ml/min/1.73m2 by CKD-Epi equation utilizing creatinine
* Fluent English-speaking
* Able to provide informed consent
* Patients with and without current tolvaptan use (prescribed by primary nephrologist) at a stable dose for ≥3 months

Exclusion Criteria:

* Estimated GFR<35 ml/min/1.73m2 (estimated from serum creatinine using the CKD-Epi equation)
* Proteinuria >500 mg/day
* Current bempedoic acid (BA) use or history of hypersensitivity to BA
* Diabetes (currently diagnosed, or fasting glucose >125 mg/dL)
* Serum uric acid >10 mg/dL or 1 or more acute gout flare within the prior year
* Known active hepatitis or abnormal baseline liver function tests (LFTs) which is defined for patients who are not taking concomitant tolvaptan as ALT, AST or direct bilirubin >1.5X ULN (upper limits of normal), or, for patients taking tolvaptan, as an ALT, AST, or direct bilirubin >ULN
* Known unstable cerebral aneurysm
* Active coronary artery disease, defined as presence of stable or unstable angina
* Systemic disease (other than hypertension) likely to contribute to kidney disease (e.g., lupus)
* Current use of simvastatin >20 mg or pravastatin >40 mg daily.
* Pregnancy or lactation
* Hemoglobin <10 g/dL
* Implanted ferromagnetic objects
* Use of an investigational product within prior 30 days or 5 half-lives, whichever is longer

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Safety as defined by rate of serious adverse events and adverse events of special interest (e.g., hyperuricemia, gout, liver transaminitis, and worsening anemia). | From enrollment to the end of treatment at 24 months
  Safety will be assessed through ascertainment of symptoms, laboratory measures, vital signs and physical exam. Serious adverse events (SAE) will be collected that occur from the time a participant signs the informed consent (at the screening visit) until the end of the study, meeting one or more of the following criteria, resulting in: 1) Resulting in death, 2) Non-elective hospitalization, 3) Life threatening (if patient continued on study drug could result in death), 4) Harming or disabling persistently or permanently , 5) Exceeding the nature, severity or frequency of risk described in the protocol, or 6) Resulting in congenital anomaly. A hepatologist with experience in drug-related liver toxicity will serve as a medical monitor. Their role is to review cases in which there is a significant elevation in liver function tests after the start of study drug and to advise on further workup, if necessary, and participant management.
Drug tolerability as assessed by the proportion of participants still taking study drug at 24 months and adherence directly measured by pill counts. | At 3, 6, 12, 18, and 24 months (at the end of treatment)
  Drug tolerability will be assessed by the proportion tolerating and taking the prescribed dose of study drug at each time point as measured by pill counts, and by a "yes" response to the question "Can you tolerate this study drug for the rest of your life?".

SECONDARY OUTCOMES:
Preliminary efficacy as assessed by changes in estimated glomerular filtration rate (eGFR) over time | At baseline, 0.5, 1.5, 3, 6, 9, 12, 15, 18, 21, and 24 months (end of study)
  We will estimate the effect of study drug on preliminary efficacy as defined by 24- month changes in eGFR decline as estimated by the CKD-Epi equations using serum creatinine and cystatin C measurements.
Preliminary efficacy as assessed by changes in the MRI-derived imaging parameter of height-adjusted total kidney volume (htTKV) over time | At baseline, 12 months and 24 months (end of study)
  We will estimate the effect of study drug on preliminary efficacy as defined by 24-month changes in height-adjusted Total Kidney Volume (htTKV) by MRI.
Health-related quality of life as assessed by the validated ADPKD-IS (Impact Scale) survey in the ADPKD population | At baseline, 3, 6, 12, 18, and 24 months (end of study)
  The ADPKD-IS survey measures the general impact of ADPKD on a patient's quality of life. Domains: Assesses physical symptoms, emotional symptoms, and fatigue. Recall Period: Last 2 weeks. Scoring: Uses a 1-5 scale, where 1 is "not at all" and 5 is "extremely".
Health-related quality of life as assessed by the validated ADPKD-PDS (Pain and Discomfort Scale) survey in the ADPKD population | At baseline, 3, 6, 12, 18, and 24 months (end of study)
  The ADPKD-PDS assesses ADPKD-related pain and discomfort in the ADPKD population. Domains: Measures different types of pain (dull kidney pain, sharp kidney pain, and fullness/discomfort) and pain's interference with daily activities. Recall Period: Last 7 days. Scoring: Uses a 1-5 scale for pain severity and interference, where 1 is "no pain" and 5 is "extreme pain".
Health-related quality of life as assessed by the validated ADPKD-UIS (Urinary Impact Scale) survey in the ADPKD population | At baseline, 3, 6, 12, 18, and 24 months (end of study)
  The ADPKD-UIS survey measures the urinary-related burden of ADPKD. Domains: Evaluates daytime urinary frequency, daytime urinary urgency, and nocturia (night-time urination). Recall Period: Last 7 days. Scoring: Uses a 1-5 scale for each item, where 1 is "not bothered at all" and 5 is "extremely bothered".

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth R Hallows, MD, PhD, FASN, Principal Investigator — University of Vermont; Stephen Seliger, MD, Principal Investigator — University of Maryland; Dana Miskulin, MD, Principal Investigator — Tufts University
Locations (3):
- United States (3):
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Tufts University Medical Center, Boston, Massachusetts
  - University of Vermont Medical Center, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Yes
All NIH and DoD applicable guidelines regarding data sharing will be followed. At the conclusion of the study, any data coded with a number will be made available to qualified individuals within the scientific community who apply for data use. The results and outcomes of the studies will be made generally available by publication with journal articles submitted to PubMed Central in compliance with NIH and other federal access guidelines.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning at the time the primary publication of results has occurred with no specific end date.
Access Criteria: At the conclusion of the study, any data coded with a number will be made available to qualified individuals within the scientific community who apply for data use through a website to be established at the time of publication of the primary study. Requests and applications for study data access will be reviewed by the BEAT-PKD Steering Committee composed of principal investigators and co-investigators of the various study sites.

REFERENCES:
- [Background] Hallows KR, Li H, Saitta B, Sepehr S, Huang P, Pham J, Wang J, Mancino V, Chung EJ, Pinkosky SL, Pastor-Soler NM. Beneficial effects of bempedoic acid treatment in polycystic kidney disease cells and mice. Front Mol Biosci. 2022 Nov 25;9:1001941. doi: 10.3389/fmolb.2022.1001941. eCollection 2022. PMID 36504724